CLINICAL TRIAL: NCT05586438
Title: Pharmacokinetics of Colistin in Critically-ill Patients With Acute Kidney Injury Who Receive Sustained Low-Efficiency Dialysis
Brief Title: Pharmacokinetics of Colistin in Critically-ill Patients With AKI Who Receive SLED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 223-2564-EC3
Record Dates: First submitted 2022-10-10; First posted 2022-10-19 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Bacterial Infections
Keywords: colistin
MeSH Terms: conditions — Bacterial Infections | interventions — colistinmethanesulfonic acid; Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- blood draws (Experimental): All patients enrolled will have PK blood samples obtained around a colistin dosing
  Interventions: Drug: Colistin Sulfomethate

INTERVENTIONS:
Drug: Colistin Sulfomethate — The patients receive colistin 150 mg intravenous once daily on non-dialysis day and receive colistin 150 mg intravenous every 12 hours on dialysis day
  Other Names: Colistin

SUMMARY:
Colistin was developed in the 1960s and preliminary pharmacokinetic studies were performed at that time. Dosing recommendations, on the basis of these pharmacokinetic studies, are listed in the drug's product information. However, there are no optimal dosing recommendations for patients with acute kidney injury who receive sustained low-efficiency dialysis. Furthermore, the science of antibiotic dosing ("pharmacodynamics") has changed significantly since the 1960s and it is quite possible that the dosing recommendations listed in the product information are not optimal. Furthermore, even though physicians refer to "colistin" administration, the only intravenous form of the drug is colistin methanesulfonate (CMS). CMS is converted in the body to colistin. Both CMS and colistin have different pharmacokinetic and antimicrobial activities. For this reason, we, the investigators at the Mahidol university, are performing a pharmacokinetic study of the intravenous CMS/colistin in patients requiring sustained low-efficiency dialysis. Plasma concentrations will be determined around a CMS/colistin dose once the drug has reached steady state. Microbiologic and clinical endpoints will be determined and will be correlated with these concentrations. The measurement of CMS and colistin levels will be determined by a laboratory in Australia.

DETAILED DESCRIPTION:
At baseline (upon signing informed consent), the following information will be collected: Demographic data - age, sex, height, weight, state of birth, underlying illnesses, underlying infection, immunosuppression, antibiotic use, laboratory results, current medication use, any other prior medical problems/history and clinical outcomes.

The research coordinator will contact the patient on days 14, 28 and 90 days after the infection to determine clinical outcome. If the patient is still an inpatient the research coordinator will visit the patient in their hospital room to evaluate the patient's health status. This visit will take about 10 minutes. If the patient has been discharged from the hospital, the patient will be contacted by telephone by the research coordinator to determine the health status, if no recent electronic medical record exists. This telephone contact will take about 10 minutes.

Blood work and microbiologic samples to be collected:

Collection of ten samples of 4 mL blood each day during two days of colistin treatment (the dialysis day and non-dialysis day) of colistin therapy will occur. These samples will be collected:

immediately pre-dose, at the end of the colistin infusion, 60 minutes after the end of the colistin infusion, 2 hours after the end of the colistin infusion, 5 hours after the end of the colistin infusion, 8 hours after the end of the colistin infusion, 12 hours after the end of the colistin infusion (or immediately prior to the next dose if the drug is being given every 12 hours).

13 hours after the end of the colistin infusion, 16 hours after the end of the colistin infusion, 20 hours after the end of the colistin infusion, 24 hours after the end of the colistin infusion, Indwelling venous and arterial access lines, if already in place, will be utilized for the pharmacological study's blood draws.

On dialysis day, collection of dialysate fluid will also occur.

60 minutes after the end of the colistin infusion, 3 hours after the end of the colistin infusion, 5 hours after the end of the colistin infusion, 7 hours after the end of the colistin infusion

Rationale: The samples will be utilized for quantification of plasma levels of colistin.

Collection of microbiologic samples within 48-96 hours of the initiation of colistin therapy. These samples are two sets of blood cultures if the patient had bacteremia, a sputum culture if the patient had pneumonia.

Rationale: These samples will be used to determine if there has been rapid bacteriologic clearance of infection.

The blood samples will be processed and stored in a -80° C freezer in a secured laboratory under the supervision of the principal investigator. These samples will then be sent to the laboratory of Drs Jian Li and Roger Nation in Melbourne, Australia, to determine the amount of colistin and CMS that reached the participant's blood following dose administration. All samples will be sent de-identified.

All samples will be analyzed to obtain the amount of colistin and CMS found in the blood. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location.

Other items to be collected for study purposes:

An unopened vial of colistin from the same batch as used for the patient will be collected for analysis, so the actual dose of colistin can be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than 18 years of age.
* All patients will remain in the hospital for pharmacokinetic sampling.
* All subjects must be on the medication colistin as part of their standard of care.
* All subjects must be on sustained low-efficiency dialysis

Exclusion Criteria:

* Pregnancy and lactation
* The patients receiving colistin inhalation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve [AUC] | 24 hours
  The area under the plasma drug concentration-time curve (AUC) reflects the actual body exposure to colistin after administration of a dose of colistin and is expressed in mg*h/L.
  Predose, and 1, 2, 5, 8, 12 hours after administration
Maximum Plasma Concentration [Cmax] | 24 hours
  Cmax is the maximum (or peak) serum concentration that colistin achieves in a specified compartment or test area of the body after colistin has been administered and before the administration of a second dose.
  Predose, and 1, 2, 5, 8, 12 hours after administration.

SECONDARY OUTCOMES:
Treatment-Related Adverse Events CTCAE v4.0 | 14 days
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Adhiratha Boonyasiri, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nation RL, Garonzik SM, Thamlikitkul V, Giamarellos-Bourboulis EJ, Forrest A, Paterson DL, Li J, Silveira FP. Dosing guidance for intravenous colistin in critically-ill patients. Clin Infect Dis. 2017 Mar 1;64(5):565-571. doi: 10.1093/cid/ciw839. Epub 2016 Dec 23. PMID 28011614
- [Background] Jitmuang A, Nation RL, Koomanachai P, Chen G, Lee HJ, Wasuwattakul S, Sritippayawan S, Li J, Thamlikitkul V, Landersdorfer CB. Extracorporeal clearance of colistin methanesulphonate and formed colistin in end-stage renal disease patients receiving intermittent haemodialysis: implications for dosing. J Antimicrob Chemother. 2015;70(6):1804-11. doi: 10.1093/jac/dkv031. Epub 2015 Feb 18. PMID 25698772